CLINICAL TRIAL: NCT03528590
Title: Ventilation Efficacy of I-gel® Size 3 and Size 4 Supraglottic Airway Devices in Anesthetized, Paralyzed Female Patients Weighing Between 50 and 60 Kilograms: a Randomized Trial
Brief Title: Ventilation Efficacy of Size 3 or Size 4 I-gel in Female Patient Weighing 50 to 60 Kilograms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201803061RIND
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Body Weight; Breast Neoplasms; Laryngeal Masks
Keywords: laryngeal mask airway; breast surgery
MeSH Terms: conditions — Body Weight; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- size 3 i-gel® (Active Comparator): size 3 i-gel supraglottic airway device in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery.
  Interventions: Device: size 3 i-gel supraglottic airway device
- size 4 i-gel® (Experimental): size 4 i-gel supraglottic airway device in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery.
  Interventions: Device: size 4 i-gel supraglottic airway device

INTERVENTIONS:
Device: size 3 i-gel supraglottic airway device — Use size 3 i-gel® in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery.
  Arms: size 3 i-gel®
Device: size 4 i-gel supraglottic airway device — Use size 4 i-gel® in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery.
  Arms: size 4 i-gel®

SUMMARY:
Currently, the main method for selecting an i-gel® size is based on the body weight recommendation (30-60 kg for size 3 and 50-90 kg for size 4) according to the manufacturer's recommendation. However, there is an overlapping in size selection in people weighing between 50 and 60 kilograms. Laryngeal mask airways are widely used for breast surgery, and this patient cohort is often weighed between 50-60 kilograms in National Taiwan University Hospital. Therefore, in this randomized clinical trial, the investigators will compare the ventilation efficacy of size 3 and size 4 i-gel® in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery. Also, the investigators will record any side effects of size 3 and size 4 i-gel® in this cohort.

DETAILED DESCRIPTION:
With the introduction of the laryngeal mask, it has been widely used for the management of airway during general anesthesia. Compared to the endotracheal tube, it has the advantages of easier and faster placing, reducing the proportion of a sore throat and other benefits. The i-gel® is a second-generation of the laryngeal mask. Compared to the classic laryngeal mask, it provides higher sealing pressure and better airway protection to reduce respiratory complications.

Choosing an appropriate size laryngeal mask is an important issue. Trauma during placing or positive ventilation failure may occur if the wrong size is selected. Currently, the main method for selecting an i-gel® size is based on the body weight recommendation (30-60 kg for size 3 and 50-90 kg for size 4) according to the manufacturer's recommendation. However, there is an overlapping in size selection in people weighing between 50 and 60 kilograms. Laryngeal mask airways are widely used for breast surgery, and this patient cohort is often weighed between 50-60 kilograms in National Taiwan University Hospital. Therefore, in this randomized clinical trial, the investigators will compare the ventilation efficacy of size 3 and size 4 i-gel® in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery. Also, the investigators will record any side effects of size 3 and size 4 i-gel® in this cohort.

Keywords: Airway management; laryngeal mask airway; breast surgery

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years old.
* ASA physical status I and II.
* Elective breast surgery.
* Female with a body weight of 50 - 60 kilograms.

Exclusion Criteria:

* High risk of aspiration. (defined as history of gastroesophageal reflux, hiatal hernia, previous gastric surgery, and those who take medications for disorders of gastrointestinal motility)
* Previous head & neck surgery.
* Previous head & neck concurrent chemoradiotherapy (CCRT)
* Reactive airway disease: chronic obstructive pulmonary disease (COPD), asthma, upper respiratory infection in recent two weeks
* Exposure to tobacco
* Pregnancy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Compare the ventilation efficacy of size 3 and size 4 i-gel® in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery. | 1 day
  Use ventilation score (1 point for presence of each item, a total score from 0 to 3) to evaluate ventilation efficacy. Ventilation score include:
  1. Air leak pressure below 15 cm H2O
  2. Bilateral chest excursion during inspiratory 20 cm H2O
  3. Square wave capnography

SECONDARY OUTCOMES:
Compare side effects of size 3 and size 4 i-gel® in anesthetized, paralyzed female patients weighing 50 to 60 kilograms who undergo breast surgery. | 2 days
  Any Side effects include:
  1. Blood stain on i-gel after removing
  2. Sore throat at post-anaesthesia care unit (PACU)
  3. Sore throat after 24 hours
  4. Dysphagia after 24 hours
  5. Mouth, lip and tongue injury
  6. Dysphonia
  7. Hiccup
  8. Myalgia

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hui Hung, MD, Principal Investigator — National Taiwan University Hospital Department of Anesthesiology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No